CLINICAL TRIAL: NCT04883190
Title: Physical and Mental Fatigue a Long COVID-19 Symptom - Substudy of FSC19-KN Trial
Brief Title: Fatigue a Long COVID-19 Symptom Substudy of FSC19-KN Trial
Acronym: SubFSC19-KN
Status: Completed | Type: Observational
Sponsor: Hegau-Bodensee-Klinikum Singen (Other)
Responsible Party: Sponsor
Other Study IDs: 21-1340
Record Dates: First submitted 2021-04-30; First posted 2021-05-12 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: SARS-CoV2 Infection
Keywords: Fatigue; Covid-19 Disease
MeSH Terms: conditions — COVID-19; Fatigue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1. after SARS-CoV-2 infection: All participants in the study and control group of the FSC19-KN study will be contacted either by email or by post.
  We plan to write to around 200-250 patients after SARS-CoV-2 infection and 200-250 test subjects in the control group.
  Interventions: Other: Fulfilling Questionaires
- 2. control group with negative antibody test: All participants in the study and control group of the FSC19-KN study will be contacted either by email or by post.
  We plan to write to around 200-250 patients after SARS-CoV-2 infection and 200-250 test subjects in the control group.
  Interventions: Other: Fulfilling Questionaires

INTERVENTIONS:
Other: Fulfilling Questionaires — Fulfilling Questionaires PHQ-D (brief) and FSMC

SUMMARY:
Prospective, controlled follow-up observation of SARS-CoV-2 positive patients with regard to the aspect of fatigue (cognitive / motor) and psychological disorders in the areas of anxiety, depression and somatization.

DETAILED DESCRIPTION:
After informed consent is given, questionnaires will be obtained 6 months and 12 months after infection. For analyzing cognitive and motor fatigue, classified in mildly, moderately or severely fatigue the questionnaire will be calculated by The Fatigue Scale for Motor and Cognitive Functions (FSMC).

And the occurrence of Major Depressive Disorder, other depressive Syndrome or Panic syndrome measured by Brief Patient Health Questionnaire.

The FSC19-KN trial already included patients with positive test for SARS-CoV-2 by PCR and volunteers with negative SARS-CoV-2 antibody testing. Verification of exclusion criteria had been completed in the main trial FSC19-KN. After the informed consent to participation in the sub-study is given all inclusion modalities are fulfilled.

ELIGIBILITY:
Inclusion Criteria:

Patient must meet ALL of the following criteria.

1. Participation in the FSC19-KN study
2. Consent to participate in the survey

Exclusion Criteria:

1. Failure to give consent to the survey

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Within the FSC19-KN trial up to 250 SARS-CoV-2 positive patients and 250 volunteers without SARS-CoV-2 infection are included.
  We plan to contact all attendees of the FSC19-KN trial which gave permission to contact via e-mail.
  They will be asked to contribute the sub-study by declaring their informed consent online. Only if their agreement of participation is given, they can fill in our online questionnaire.
Sampling Method: Non-Probability Sample
Enrollment: 353 (Actual)
Dates: Start 2021-05-15 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Presence of fatigue | 6 month after infection
  Evaluate cognitive and motor fatigue classified in mildly, moderately or severely fatigue
Presence of fatigue | 12 month after infection
  Evaluate cognitive and motor fatigue classified in mildly, moderately or severely fatigue

SECONDARY OUTCOMES:
Occurrence of Major Depressive Disorder, other depressive Syndrome or Panic syndrome. | 6 month after infection
  analyzed by PHQ-D (brief)
Occurrence of Major Depressive Disorder, other depressive Syndrome or Panic syndrome. | 12 month after infection
  analyzed by PHQ-D (brief)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Kollum, PD Dr., Principal Investigator — Hegau-Bodensee-Klinikum Singen
Locations (1):
- Hegau Bodensee Klinikum Singen, Singen, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No
The aim is to publish the results in a peer reviewed medical journal without sharing any participant data

REFERENCES:
- [Result] Sabrina Geng, Jonas Haberland, Elisabeth Haberland, Julia Hromek, Heidi Zimmermann, et al, (2024), Effects on Fatigue and Depression 11 And 19 Months after a Sars-Cov-2 Infection a Case Control Study, J. Clinical Cardiology and Cardiovascular Interventions, 7(2); DOI:10.31579/2641-0419/348